CLINICAL TRIAL: NCT05626166
Title: Clinical Study Evaluating the Efficacy and Safety of Diosmin in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: the Efficacy and Safety of Diosmin in Patients With Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amira B ismail, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36031/11/22
Record Dates: First submitted 2022-11-09; First posted 2022-11-23 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Diosmin

STUDY DESIGN:
Intervention Model Description: This proof of concept study will be designed to be a randomized, double-blind, placebo controlled parallel study. The study will be conducted on 60 patients with mild to moderate ulcerative colitis receiving mesalamine. Patients will be recruited from Tropical Medicine Department, Tanta University Hospital, Tanta, Egypt. The patient will be followed for 3 months. The blindness will be maintained by the similarity in appearance, color and shape between placebo and diosmin tablets. The patients will be randomized in a 1:1 ratio by neutral researcher using sealed envelopes methods with assignment codes into the following two groups: Group I (Control group; n=30) which will receive mesalamine 1000 mg three times daily plus placebo tablets twice daily for 3 months.
  Group II: (Diosmin group; n=30) which will receive mesalamine 1000 mg three times daily plus diosmin 600 mg twice daily for 3 months
Who Masked: Participant, Investigator
Masking Description: This proof of concept study will be designed to be a randomized, double-blind, placebo controlled parallel study, The blindness will be maintained by the similarity in appearance, color and shape between placebo and diosmin tablets.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Group I (Control group; n=30) which will receive mesalamine 1000 mg three times daily plus placebo tablets twice daily for 3 months.
  Interventions: Drug: Placebo
- diosmin group (Experimental): Group II: (Diosmin group; n=30) which will receive mesalamine 1000 mg three times daily plus diosmin 600 mg twice daily for 3 months.
  Interventions: Drug: Diosmin

INTERVENTIONS:
Drug: Placebo — placebo tablets twice daily
  Arms: control group
Drug: Diosmin — diosmin 600 mg twice daily
  Other Names: diosimax
  Arms: diosmin group

SUMMARY:
This is a randomized, controlled study evaluating diosmin tablets administered daily for 3 months. The purpose of the study is to evaluate the efficacy and safety of diosmin in the treatment of mild to moderately active ulcerative colitis. Disease activity will be measured using modified truelove and witt's classification.

DETAILED DESCRIPTION:
This study aims at evaluating the efficacy and safety of diosmin as add-on therapy to mesalamine in patients with mild to moderate ulcerative colitis.

This proof of concept study will be designed to be a randomized, double-blind, placebo controlled parallel study. The study will be conducted on 60 patients with mild to moderate ulcerative colitis receiving mesalamine. The patient will be followed for 3 months.

The patients will be randomised into the following two groups:

Group I (Control group; n=30) which will receive mesalamine 1000 mg three times daily plus placebo tablets twice daily for 3 months.

Group II: (Diosmin group; n=30) which will receive mesalamine 1000 mg three times daily plus diosmin 600 mg twice daily for 3 months.

All participants included in this study will be subjected to the following:

1. Demography, history, and physical examination
2. Blood sample collection and biochemical assessment At baseline and after the intervention, 10 ml of venous blood will be withdrawn from each participant.

3 ml of blood will be used for immediate determination of routine parameters including:

* Hemoglobin concentration.
* Ertherythrocyte sedimentation rate (ESR).
* Prothrombin time.

Two ml of blood will be immediately centrifuged at 3000 rpm for 10 min for immediate determination of:

- Serum albumin

The remaining 5 ml of blood will be used for the analysis of the biological parameters which include:

* Malondialdehyde (MDA) as oxidative stress marker (colorimetry).
* Tumor necrosis factor-alpha (TNF-α) as pro inflammatory marker (ELISA).
* Caspase-3 as a potential marker for apoptosis (ELISA). 3. Clinical assessment

Clinical assessment will be done through determination of:

A. Disease severity which will be assessed according to the modified Truelove and Witt's classification.

B. The activity index (AI) for ulcerative colitis which is expressed as follows:

AI = 60 x blood stool + 13 x bowel movements (frequency of defection) + 0.5 x ESR - 4 x Hb - 15 x albumin + 200.

C. Health-related Quality of Life (HRQoL) using The Short Inflammatory Bowel Disease Questionnaire (SIBDQ).

D. Assessement of pain score through the brief pain inventory short form "BPI-SF" worst item.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old.
* Both male and female sex.
* Newly diagnosed patients with mild and moderate ulcerative colitis and treated with 5-aminosalicylic acid (mesalamine).

Exclusion Criteria:

* Patients with severe ulcerative colitis.
* Patients with colorectal cancer.
* Patients on rectal or systemic steroids.
* Patients on immunosuppressants or biological therapies.
* Patients with previously failed treatment with sulphasalazine.
* Patients with known allergy to study medications.
* History of complete or partial colectomy.
* Patients with heart diseases and arrhythmia.
* Patients on blood thinning agents.
* Patients on anticoagulants (warfarin), anticonvulsants (carbamazepine and phenytoin), muscle relaxants (chlorzoxazone) and non-steroidal anti-inflammatory drugs (diclofenac).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
the change in Truelove and Witt's classification. | at baseline then after 3 months
the change in health related quality of life (HRQoL) questionnaire | at baseline then after 3 months

SECONDARY OUTCOMES:
the change in the measured biological parameters (TNF alpha, MDA, caspase-3) | at baseline then after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: tarek M mostafa, professor, Principal Investigator — Tanta University
Locations (1):
- Tanta university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No